CLINICAL TRIAL: NCT06141161
Title: Assessment of Bronchial Asthma Among Patients Attending Sohag University Hospital
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Doha Mohamed Ismail, Resident of chest department, Sohag university hospital, Sohag University
Other Study IDs: Soh-Med-23-10-015MS
Record Dates: First submitted 2023-11-15; First posted 2023-11-21 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Bronchial Asthma
MeSH Terms: conditions — Asthma | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group A,: group A (controlled bronchial asthma patients)
  Interventions: Drug: corticosteroids
- group B: group B(uncontrolled bronchial asthma patients)
  Interventions: Drug: corticosteroids

INTERVENTIONS:
Drug: corticosteroids — inhailed or oral corticosteroids

SUMMARY:
Asthma is a significant public health threat, affecting more than 300 million individuals globally. Asthma is classified as a non-communicable disease and leads to reduced quality of life, poor physical functioning and reduced emotional well-being. The impact of this disease can be widespread and extends beyond the person living with the disease, affecting the lives of their family members, carers, communities and the health care system (1).

Asthma is a variable chronic respiratory condition. It is characterized by symptoms of wheeze, cough, chest tightness, dyspnea and backed by variable airflow limitation, airway inflammation and airway hyper-responsiveness (AHR). The severity of asthma varies considerably, both between individuals and within individuals over time. Some people may have intermittent asthma and others may experience severe, potentially life-threatening disease (2, 3,4).

ELIGIBILITY:
Inclusion Criteria:

* bronchial asthma patients aged more than 18 years, both sexes are included

Exclusion Criteria:

* children ,patients who are unable to do spiromerty or contrindecated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: bronchial asthma patients aged more than 18 years of both sexes
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
percent of controlled bronchial asthma patients | 12 months
  to detect percent of controlled patients

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University hospitals, Sohag, Egypt

REFERENCES:
- [Background] Dashash NA, Mukhtar SH. Prescribing for asthmatic children in primary care. Are we following guidelines? Saudi Med J. 2003 May;24(5):507-11. PMID 12847627
- [Background] Al-Moamary MS, Alhaider SA, Al-Hajjaj MS, Al-Ghobain MO, Idrees MM, Zeitouni MO, Al-Harbi AS, Al Dabbagh MM, Al-Matar H, Alorainy HS. The Saudi initiative for asthma - 2012 update: Guidelines for the diagnosis and management of asthma in adults and children. Ann Thorac Med. 2012 Oct;7(4):175-204. doi: 10.4103/1817-1737.102166. PMID 23189095
- [Background] Braido F, Canonica GW. Worldwide differences on the concept of control of asthma. Ther Adv Respir Dis. 2008 Feb;2(1):3-5. doi: 10.1177/1753465807087091. PMID 19124353
- [Background] National Asthma Education and Prevention Program. Expert Panel Report 3 (EPR-3): Guidelines for the Diagnosis and Management of Asthma-Summary Report 2007. J Allergy Clin Immunol. 2007 Nov;120(5 Suppl):S94-138. doi: 10.1016/j.jaci.2007.09.043. PMID 17983880